CLINICAL TRIAL: NCT07074626
Title: Efficacy of Local Lidocaine Gel for Pain Management During Transrectal Sonography in Virgins With Suspected Pelvic Pathology, A Phase II Single Arm Interventional Study
Brief Title: Local Lidocaine Gel for Pain Management During
Status: Active, not recruiting | Type: Observational
Sponsor: Suez University (Other)
Responsible Party: Principal Investigator, Ahmed Sewidan, lecturer, Suez University
Other Study IDs: 2
Record Dates: First submitted 2025-07-06; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Ultrasound Diagnostics
Keywords: transrectal ultrasound
MeSH Terms: interventions — Ultrasound, High-Intensity Focused, Transrectal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: A 45 virgin attending Suez university hospital gynecology outpatient clinic for collection of baseline data, including demographic information, medical history, body mass index (BMI).
  Interventions: Other: transrectal ultrasound

INTERVENTIONS:
Other: transrectal ultrasound — A- Complete history was taking (personal, past, medical, surgical and family history) with careful attention to abdominal examination and suspected cause of pelvic pathology B- Through physical examination (general and abdominal examination). C- Investigations.
  * Trans-rectal ultrasound will be conducted to all the virgin patients as the standard US examination to detect the pelvic pathology
  * Patient anticipation for pain will be documented before the exam according to pain visual analogue scale (VAS)
  * Lidocaine gel will be used on the probe during TRU
  * The intensity of pain during trans-rectal US based on the pain visual analogue scale (0-10 ) points and the adverse events like extreme pain, inability to complete the examination and inability to detect the pathology will be reported.A Visual Analogue Scale (VAS) is one of the valided pain rating scales used for the first time in 1921 by Hayes and Patterson.

SUMMARY:
Ultrasound is a very useful diagnostic tool in the obstetrics and gynecologic field. It is used to diagnose pelvic organs including the uterus, ovaries, tubes and endometrium, and can be used to evaluate gynecologic tumors regardless of their risk of malignant index. The types of pelvic sonography according to route include transvaginal sonography (TVS), transabdominal sonography (TAS), and transrectal sonography (TRS). Insertion of the probe into the vagina allows a very close and clear view of the pelvic organs, physicians have preferred TVS to TAS for accurate diagnosis of pelvic pathology .

DETAILED DESCRIPTION:
TVS is not acceptable because of a virginal introitus, agenesis of the vagina, or patient refusal of the introduction of a probe into the vagina, TRS may be a useful alternative tool for evaluating pelvic organs. The rectal administration of a local anesthetic, lidocaine gel, was recently proposed to reduce the pain of TRS-guided biopsy of the prostate. A similar result was also shown in a study evaluating the efficacy of lidocaine gel in rigid cystoscopy. However, data on the efficacy of lidocaine gel on providing the pain relief during TRS in gynecologic patients are lacking. Considering the clinical situation that many women have hesitated to undergo TRS because of concerns about pain, studies investigating methods for relieving pain during TRS are needed.

Recently, there are different type of scale, that are used for assessing pain but without any valid (accurate) and reliable (reproducible) instruments it is difficult to have real effect of treatment. The most commonly used pain scales are the Visual Analogue Scale (VAS), the Numerical Rating Scale (NRS) the Verbal Rating Scale (VRS) .

VAS is used in epidemiological and clinical research to calculate the intensity and frequency of a variety of clinical symptoms. In randomized controlled trials (RCT) and clinical trials (CT) VAS is frequently used to determine the effectiveness of treatment as an outcome measure. VAS is also very much popular in the gynecological area. In post operative pain assessment this scale is applied to measure pain. Moreover, after caesarean section the VAS is used to assessing pain

ELIGIBILITY:
Inclusion Criteria:

* Virgins
* Patients with undiagnosed acute pelvic pain
* Patients with undiagnosed abnormal uterine bleeding
* Parents consent for patients less than 18 years

Exclusion Criteria:

* Medical history of allergy to lidocaine
* Chronic pelvic pain
* Chronic pain condition for which patients were taking daily pain medication
* Anorectal pathologies

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: virgins attending the clinic with suspected pelvic pathology
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Decrease the intensity of pain associated with lidocaine gel during trans-rectal ultrasound in compraison with patients exepectaions before the TRU examination by using Visual Analogue Scale, which is one of the valided pain rating scales. | 3 months
  A Visual Analogue Scale is one of the valided pain rating scales used for the first time in 1921 by Hayes and Patterson.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed ElSherbiny, Principal Investigator — faculty of medicine, Suez university Suez, Suez, Egypt
Locations (1):
- faculty of medicine, Suez university, Suez, Suez Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Background] Nam SH, Kim KH, Choi C, Nam SH, Song T, Lee KW. Lidocaine gel versus plain lubricating gel for pain reduction during transrectal sonography (LIPS): A randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2017 May;212:60-64. doi: 10.1016/j.ejogrb.2017.03.012. Epub 2017 Mar 11. PMID 28342390
- [Background] Begum MR, Hossain MA. Validity and reliability of visual analogue scale (VAS) for pain measurement. Journal of Medical Case Reports and Reviews. 2019;2(11).
- [Background] Stourac P, Kucharova E, Krikava I, Maly R, Kosinova M, Harazim H, Smekalova O, Bartikova I, Stoudek R, Janku P, Huser M, Wagnerova K, Haklova O, Hakl L, Schwarz D, Zelinkova H, Littnerova S, Jarkovsky J, Gal R, Sevcik P. Establishment and evaluation of a post caesarean acute pain service in a perinatological center:retrospective observational study. Ceska Gynekol. 2014 Nov;79(5):363-70. PMID 25472454
- [Background] Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, Fainsinger R, Aass N, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011 Jun;41(6):1073-93. doi: 10.1016/j.jpainsymman.2010.08.016. PMID 21621130
- [Background] Goktug HN, Ozturk U, Sener NC, Tuygun C, Bakirtas H, Imamoglu MA. Do lubricants with 2% lidocaine gel have an effect on patient comfort in diagnostic cystoscopy? Adv Clin Exp Med. 2014 Jul-Aug;23(4):585-7. doi: 10.17219/acem/37229. PMID 25166443
- [Background] Irani J, Fournier F, Bon D, Gremmo E, Dore B, Aubert J. Patient tolerance of transrectal ultrasound-guided biopsy of the prostate. Br J Urol. 1997 Apr;79(4):608-10. doi: 10.1046/j.1464-410x.1997.00120.x. PMID 9126093
- [Background] Renfer LG, Vaccaro JA, Kiesling V. Digital-directed transrectal core biopsy with spring-loaded biopsy device (Biopty). Urology. 1991 Aug;38(2):161-2. doi: 10.1016/s0090-4295(05)80079-2. No abstract available. PMID 1877135
- [Background] Qureshi IA, Ullah H, Akram MH, Ashfaq S, Nayyar S. Transvaginal versus transabdominal sonography in the evaluation of pelvic pathology. J Coll Physicians Surg Pak. 2004 Jul;14(7):390-3. PMID 15279738
- [Background] Park JW, Hwang SO, Park JH, Lee BI, Lee JH, Kim KW, et al. Discrimination between Benign and Malignant Pelvic Masses Using the Risk of Malignancy Index 1. J Korean Soc Menopause. 2013;19:18-25.